CLINICAL TRIAL: NCT06796023
Title: Comparison Between Lumbar Stabilization Exercises and Lumbar Manipulation on Multifidus Muscle in Chronic Low Back Pain: Randomized Control Trial
Brief Title: Comparison Between Lumbar Stabilization Exercises and Lumbar Manipulation on Multifidus Muscle in Chronic Low Back Pain This Study Will Investigate and Compare the Effect of Lumbar Stabilization Exercises and Manipulation on Multifidus Muscle in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas Abutaleb, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004972
Record Dates: First submitted 2025-01-11; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Chronic Low Back Pain (CLBP)
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stretching and strengthening exercises (Active Comparator): Stretching and strengthening exercises for back muscles
  Interventions: Other: Stretching and strengthening exercises for back muscles
- Lumbar Stabilization (Experimental): Lumbar Stabilization exercises
  Interventions: Other: Stretching and strengthening exercises for back muscles; Other: Lumbar stabilization Exercises
- Lumbar Manipulation (Experimental): Lumbar Manipulation
  Interventions: Other: Stretching and strengthening exercises for back muscles; Other: Lumbar Manipulation

INTERVENTIONS:
Other: Stretching and strengthening exercises for back muscles — Stretching and strengthening exercises for back muscles
Other: Lumbar stabilization Exercises — Lumbar stabilization Exercises
  Arms: Lumbar Stabilization
Other: Lumbar Manipulation — Lumbar Manipulation
  Arms: Lumbar Manipulation

SUMMARY:
Histological and morphological changes of multifidus muscle have been reported in lumbar disc herniation (LDH), but there is scarce research comparing the efficacy of different treatment programs that can correct multifidus dysfunction in chronic low back pain (LBP) with LDH. The purpose: this study will be to investigate and compare the effect of lumbar stabilization exercises and manipulation on multifidus muscle in chronic LBP patients with LDH. Subjects: sixty patients aged ranged from 45 - 65 years suffering from chronic LBP with LDH will be randomly assigned into three groups, each group includes 20 patients. Method: group (A) (control group) will receive general exercises for back muscles, group (B) will receive general exercises and lumbar stabilization exercises, and group (C) will receive general exercises and lumbar manipulation (B and C experimental groups). The outcome measurements pre and post 6 weeks of treatment will be pain intensity by visual analogue scale (VAS), functional disabilities by Oswestry disability index (ODI), lumbar repositioning by Biodex system (LR), cross sectional area (CSA) and the asymmetry of both sides of multifidus muscle at the fourth and fifth lumbar vertebrae by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* The selected subjects had chronic LBP with magnetic resonance imaging (MRI) evidence of disc herniation at levels of L4-L5 and/or L5-S1 diagnosed by physician (orthopedist, neurosurgeon).
* A period of continuous complaints of pain for more than 12 weeks.
* All patients reported an average pain level of at least 5 on a scale of 0 to 10.

Exclusion Criteria:

* Acute inflammatory diseases of musculoskeletal system.
* Pathology or deformities of hip, knee and ankle joints.
* History of surgical approach to their back or had special pathology or non spinal condition causing referred back symptoms.
* Patient who indicated for surgery to treat lumbar disc herniation (i.e. sever intolerable pain, motor weakness, and cannot control urine and stool).
* Cardiopulmonary diseases which decrease the patient's tolerance and activities.
* Spondylolisthesis.
* Diabetic neuropathy.
* Osteoporosis.
* A recent history of vestibular disorder or inner ear infection with associated balance and coordination problems.
* A history of cerebral trauma with unresolved neurosensory symptoms or neurological deficits.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | pre and post 6 weeks
  The patients will asked about the perception of pain using a 10 cm line with 0 (no pain) on one end and 10 (worst pain) on the other end. Patients will be asked to place a mark along the line to dente their level of pain.
functional disabilities by Oswestry disability index | pre and post 6 weeks
  It consists of 10 multiple- choice questions of back pain included disability in daily function and leisure time activities, for each question the patient selects one sentence out of six that best described his disability. For each section of six statements the total score is 5; if the first statement is marked, the score is zero, if the last is marked the score is 5. The final score calculated as follow:
  Total score\ (5 x number of questions answered) x 100%. The maximal score is 50 (maximum disability) and the result taken as a percentage from the total score. High score indicate greater disability. Score from 0 to20% indicate minimal disability, score from 20 to 40% indicate moderate disability, score from 40 to 60% indicate sever disability, score from 60 to80% indicate crippled disability, and score from 80 to 100% indicate that the patient confined to bed
lumbar repositioning angle | pre and post 6 weeks
  Biodex system 3 pro Isokinetic dynamometer (Biodex Medical INC., Shirley, New York, USA), equipped with a special forward reclined back attachment, will be used to measure the lumbar repositioning angle of the lumbar region.
  * The participant will be positioned in 30° of lumbar flexion for 10 seconds and then instructed to remember the position because he/she will be asked to reproduce this position.
  * The participant returns to the neutral position and then will be given the verbal instruction of reproducing the target position as accurately as he/she could.
  * The subject will hold the final position for 3 seconds. The test will be repeated 3 times. The mean deviation or absolute error about the 30° target position will be calculated each time.
Cross sectional area of multifidus muscle | pre and post 6 weeks
  Ultrasonography instrument (Phillips HDI 5000) with a frequency 3.5-5 MHz will be used to measure the cross sectional area of multifidus muscles at levels of Lumbar vertebrae (4) and Lumbar vertebrae (5)

IPD SHARING:
Plan to Share IPD: No